CLINICAL TRIAL: NCT04797897
Title: A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in Unicondylar Knee Arthroplasty (UKA) Procedures
Brief Title: Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in Unicondylar Knee Arthroplasty (UKA) Procedures
Acronym: CORI RCT UKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study terminated prematurely due to very low patient enrollment in the study.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORI.2019.06
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Non-inflammatory Degenerative Joint Disease; Osteoarthritis; Avascular Necrosis; Requires Correction of Functional Deformity; Fracture, Knee
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Knee Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CORI UKA (Experimental): Subjects in need for unicondylar knee arthroplasty (UKA) as decided by their doctor and treated with CORI.
  Interventions: Device: CORI
- Conventional UKA (Active Comparator): Subjects in need for unicondylar knee arthroplasty (UKA) as decided by their doctor and treated with conventional approach with conventional manual instrumentation.
  Interventions: Device: Conventional

INTERVENTIONS:
Device: CORI — unicondylar knee arthroplasty (UKA) treated with CORI
  Arms: CORI UKA
Device: Conventional — unicondylar knee arthroplasty (UKA) treated with conventional approach with conventional manual instrumentation
  Arms: Conventional UKA

SUMMARY:
This is a prospective study to demonstrate the safety and effectiveness of CORI and to register CORI in China mainland.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized study to demonstrate the safety and effectiveness of CORI. In addition, the study will support regulatory approval by the National Medical Products Administration (NMPA) in China.

The study will have two arms, the investigational group will be total knee arthroplasty (TKA) using CORI, the comparison group will be conventional approach with conventional manual instrumentation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a suitable candidate for a UKA procedure using CORI and a compatible S+N Knee implant system.
2. Subject requires a cemented UKA as a primary indication that meets any of the following conditions:

   1. Non-inflammatory degenerative joint disease, including osteoarthritis
   2. Avascular necrosis
   3. Requires correction of functional deformity
   4. Requires treatment of fractures that were unmanageable using other techniques
3. Subject is of legal age to consent and considered skeletally mature (≥ 18 years of age at the time of surgery).
4. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethics Committee (EC) or Institutional Review Board (IRB) approved informed consent form.
5. Subject plans to be available through one (1) year postoperative follow-up.
6. Applicable routine radiographic assessment if possible.

Exclusion Criteria:

1. Subject receives a UKA on the index joint as a revision for a previously failed surgery, or need for complex implants, or any other implant than a standard UKA (e.g. stems, augments, or custom made devices).
2. Subject has been diagnosed with post-traumatic arthritis
3. Subject receives simultaneous bilateral UKA OR a unilateral UKA with contralateral TKA.
4. Subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator:-Contralateral primary TKA or UKA, however, the subject can only have one knee enrolled in this study.
5. Subject does not understand the language used in the Informed Consent Form.
6. Subject does not meet the indication or is contraindicated for UKA according to specific S+N knee system's Instructions For Use (IFU).
7. Subject has active infection or sepsis (treated or untreated).
8. Subject is morbidly obese with a body mass index (BMI) greater than 40.
9. Subject is pregnant or breast feeding at the time of surgery.
10. Subject, in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and was better suited for an alternate procedure.
11. Subject currently enrolled in another orthopedic clinical trial study.
12. Subject has a condition(s) that may interfere with the UKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
13. Subject in the opinion of the Investigator has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, intellectual disability, drug or alcohol abuse.
14. Subject, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.
15. Subject is a prisoner or meets the definition of a Vulnerable Subject per ISO 14155:2020 Section 3.55.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia McCracken, Study Director — Smith & Nephew, Inc.
Locations (3):
- Northern Hospital, Epping, Australia
- The Prince of Wales Hospital, Shatin, Hong Kong
- North Shore Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 4 participants enrolled & randomized into the study with each contributing one study knee.
Period: Overall Study
Arm/Group | CORI UKA | Conventional UKA
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Study Termination by Sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CORI UKA | Conventional UKA | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 1 | 2
  Hong Kong | 1 | 0 | 1
  Australia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Leg Alignment
Description: The number of participants with knees achieving post-operative leg alignment was taken by radiographic assessment at 6 weeks. Post-operative leg alignment was achieved when the deviation from the participant specific target did not exceed ±3 degrees.
Time Frame: 6 weeks
Population: Overall number of participants analyzed included those enrolled in the study with data collected for the outcome and time frame specified. Leg alignment not collected for 1 participant in CORI UKA group, and target data was not collected for 1 participant in Conventional UKA group.
Measure: Count of Participants; unit: Participants
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

2. Secondary Outcome: Component Alignment: Femoral Antero-Posterior (A/P) Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. From the A/P radiograph, the femoral flexion angle in degrees was obtained using standard radiographic tools. Femoral flexion angle is defined as the angle formed between a line across the base of the femoral condyles and a line that is centered along the femoral canal.
Time Frame: 6 weeks
Population: Overall number of participants analyzed included those enrolled with data collected for the outcome and time frame specified.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 1 | 2
degrees | 97 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 95 (1.41)

3. Secondary Outcome: Component Alignment: Tibial Antero-Posterior (A/P) Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. From the A/P radiograph, the tibial angle denotes the angle formed on the medial side of the knee from intersecting lines parallel to the tibial base plate and a line drawn parallel to the tibial canal.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 1 | 2
degrees | 84 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 89 (5.66)

4. Secondary Outcome: Component Alignment: Total Antero-Posterior (A/P) Valgus Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. The total valgus angle is the sum of the femoral flexion angle and the tibial angle.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 1 | 2
degrees | 181 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 184 (7.07)

5. Secondary Outcome: Component Alignment: Lateral View Femoral Flexion Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. The lateral view femoral flexion angle in degrees was obtained from the intersection of a line from the center of the femoral implant to the top of the femur with a line through the femoral canal. The angle is measured on the proximal side of the intersection.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 1 | 2
degrees | 0 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 5 (0)

6. Secondary Outcome: Component Alignment: Lateral View Tibial Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. The lateral view tibial angle in degrees was obtained from the intersection of a line drawn parallel to the bottom of the tibial base insert and a line through the center of the tibial base and the tibial canal.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 1 | 2
degrees | 86 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 85.5 (0.71)

7. Secondary Outcome: Radiographic Assessment
Description: Radiographic assessment measured by number of participants with any radiographic finds on antero-posterior (A/P) and lateral (L) views (yes/no). Radiographic findings indicated the presence of radiolucent lines, osteolysis & implant migration.
Time Frame: 12 months
Population: Overall number of participants analyzed indicated those enrolled in the study with data collected for the outcome and time frame specified. Data was not collected for 2 participants due to the early termination of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 1 | 1
Participants
  No | 1 | 1
  Yes | 0 | 0

8. Secondary Outcome: 2011 Knee Society Score (KSS): Objective Knee Score
Description: The 2011 Knee Society Score consists of 4 separate sub-scales. The "Objective" Knee Score is seven items with a range of 0 to 100, with a higher score indicating a better outcome.
Time Frame: Baseline, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 49 (32.53) | 33.5 (3.54)
  6 weeks | 62.5 (4.95) | 57 (7.07)
  6 months | 61.5 (4.95) | 50.5 (17.68)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 70 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 49 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

9. Secondary Outcome: 2011 Knee Society Score (KSS): Satisfaction Knee Score
Description: The 2011 Knee Society Score consists of 4 separate sub-scales. The Patient Satisfaction Score is five items with a range of 0 to 40, with a higher score indicating a better outcome.
Time Frame: Baseline, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 19 (1.41) | 10 (2.83)
  6 weeks | 24 (0) | 23 (4.24)
  6 months | 28 (2.83) | 26 (2.83)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 34 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 30 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

10. Secondary Outcome: 2011 Knee Society Score (KSS): Expectation Score
Description: The 2011 Knee Society Score consists of 4 separate sub-scales. The Patient Expectation Score is three items with a range of 0 to 15, with a higher score indicating a better outcome. The Expectation score indicates the patient's opinion on the extent they expect the operation to improve their knee pain, and ability to perform activities of daily living and recreational activities.
Time Frame: Baseline, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 13 (1.41) | 11 (1.41)
  6 weeks | 9.5 (3.54) | 8.5 (3.54)
  6 months | 11 (5.66) | 10 (1.41)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 8 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 9 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

11. Secondary Outcome: 2011 Knee Society Score (KSS): Functional Score
Description: The 2011 Knee Society Score consists of 4 separate sub-scales. The Functional Score is nineteen items with a range of 0 to 100, with a higher score indicating a better outcome. Functional Score is derived from assessments of walking and standing, standard activities, advanced activities, and discretionary activities.
Time Frame: Baseline, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 30 (11.31) | 35.5 (4.95)
  6 weeks | 37.5 (16.26) | 52 (19.80)
  6 months | 59 (7.07) | 72.5 (2.12)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 60 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 83 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

12. Secondary Outcome: Oxford Knee Score (OKS)
Description: The Oxford Knee Score (OKS) is a Patient Reported Outcome questionnaire that was developed to assess perceived function and pain answered on a Likert scale. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.
Time Frame: Baseline, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 22.5 (0.71) | 18.5 (3.54)
  6 weeks | 16 (2.83) | 29.5 (2.12)
  6 months | 35.5 (0.71) | 35 (8.49)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 38 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 41 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

13. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The Forgotten Joint Score (FJS) comprises measures for the assessment of joint-specific patient reported outcomes. Participants are asked to rate their awareness of their knee arthroplasty in 12 questions with a five point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living (i.e., a higher score is a better outcome).
Time Frame: 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  6 weeks | 13.54 (10.31) | 29.17 (11.79)
  6 months | 52.08 (8.84) | 67.71 (1.47)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 18.75 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 87.5 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

14. Secondary Outcome: Five-level EuroQol Five-dimensional (EQ-5D-5L): Index Score
Description: The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale (VAS). The descriptive system (i.e., index score) is used to describe the participant's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate their health state by marking the most appropriate statement in each of the five areas. The EQ-5D-5L Index Score was based on a scale of 0 to 1, with higher index values indicating better health and lower index values indicating worse health.
Time Frame: Baseline, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 0.71 (0.03) | 0.58 (0.01)
  6 weeks | 0.69 (0.13) | 0.79 (0.01)
  6 months | 0.81 (0.02) | 0.83 (0.04)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 0.80 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 0.77 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

15. Secondary Outcome: Five-level EuroQol Five-dimensional (EQ-5D-5L): Visal Analogue Scale (VAS) Score
Description: The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale (VAS). The VAS records the participant's self-rated health on a vertical visual analogue scale. The scale ranges from 0 to 100 where 0 indicates 'The worst health you can imagine' and 100 indicates 'The best health you can imagine'.
Time Frame: Baseline, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI UKA | Conventional UKA
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 67.5 (17.68) | 55 (7.07)
  6 weeks | 72.5 (10.61) | 72.5 (10.61)
  6 months | 85 (7.07) | 72.5 (17.68)
  12 months: number analyzed (Participants) | 1 | 1
  12 months | 80 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 75 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected from procedure to study termination, approximately 12 months.
Arm/Group | CORI UKA | Conventional UKA
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CORI UKA (N=2) | Conventional UKA (N=2)
BROKEN ANKLE (Musculoskeletal and connective tissue disorders) | 1 | 0 — Unrelated to device & procedure
INCREASED PAIN AND SWELLING IN RIGHT LEG (Musculoskeletal and connective tissue disorders) | 0 | 1 — Unrelated to device & procedure
BILATERAL PULMONARY EMBOLISM (PE) & DEEP VEIN THROMBOSIS (DVT) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Unrelated to device & procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CORI UKA (N=2) | Conventional UKA (N=2)
RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Unrelated to device & procedure
PAIN IN KNEE, PREPATELLAR SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0 — Unrelated to device, possible relationship to procedure
BURNING AND ALTERED SENSATION AROUND LATERAL ASPECT OF SURGICAL WOUND. (General disorders) | 1 | 0 — Unrelated to device & procedure
POSSIBLE PARKINSON'S (Nervous system disorders) | 0 | 1 — Unrelated to device & procedure

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to low enrollment leading to a small number of participants analyzed. Meaning or reliable results could not be determined from the limited data available from 4 participants because of the early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period up to 40 days but less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor may request removal of specified Confidential Information (other than results of the study) to the communication as is reasonably required to protect the Intellectual Property of the sponsor and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04797897/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04797897/SAP_001.pdf